CLINICAL TRIAL: NCT02230111
Title: Impact of Cognitive Dietary Restraint on Perceived Stress, Appetite Sensations and Food Cravings During Energy Restriction in Women With Obesity
Brief Title: Impact of Cognitive Dietary Restraint on Perceived Stress, Appetite Sensations, Food Cravings During Energy Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Principal Investigator, Simone Lemieux, Professor, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-170
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Overweight
Keywords: Women; Caloric restriction; Cognitive dietary restraint; Eating behaviours; Food habits; Appetite sensations; Stress; Weight management
MeSH Terms: conditions — Overweight; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy restriction plus CDR group (Experimental): Subjects will receive a reduced-calorie low energy density diet which will provide 85% of their energy needs for a period of 4 weeks. They will be told that they are on a low-calorie diet and strategies to increase CDR will be used.
  Interventions: Behavioral: Energy restriction plus CDR
- Energy restriction without CDR group (Experimental): Subjects will receive a reduced-calorie low energy density diet which will provide 85% of their energy needs for a period of 4 weeks. To have a condition of energy restriction without CDR, they will not be told that they are on a low-calorie diet and non-restrictive messages will be used.
  Interventions: Behavioral: Energy restriction without CDR

INTERVENTIONS:
Behavioral: Energy restriction plus CDR — Subjects will receive a reduced-calorie low energy density diet which will provide 85% of their energy needs for a period of 4 weeks. In the condition in which an increase in CDR will be induced, women will be told at the beginning of the study and will be reminded throughout the 4-week duration of the experimental condition that they are on a low-calorie diet and that it is important not to eat more than what is provided and that they should strictly avoid non-study food if they want to lose weight and improve their blood pressure. Subjects will receive feedback about their weight trajectory. After the 4-week controlled intervention women will then receive further information and advices to pursue their weight loss on their own and keeping on with strategies relying on an increase in CDR.
  Arms: Energy restriction plus CDR group
Behavioral: Energy restriction without CDR — Subjects will receive the same low-calorie diet (85% of their energy needs) for 4 weeks but will not be told that they are on an energy-deficit diet. They will be told at the beginning of the study that the food provided cover all their nutrient needs and that they should eat until satiation. There will be no emphasis on body weight and subjects will be reminded that the aim of the intervention is to document the effects of a diet rich in vegetables and fruits on blood pressure. After the 4-week controlled diet, participants will be taught about the impact of a low energy density diet on satiation and satiety. They will receive further information and advices (with non-restrictive messages) to incorporate more vegetables and fruits in their usual diet.
  Arms: Energy restriction without CDR group

SUMMARY:
The purpose of this study is to measure the effects of a reduced-calorie low energy density diet with and without increased cognitive dietary restraint (CDR) on stress (biological markers and perceived stress), eating behaviours, appetite sensations, anthropometric variables and women's attitude toward their children's eating behaviours in premenopausal overweight/obese women in both the short term (immediately after the end of the 4-week intervention) and longer term (3 months after the end of the intervention). The investigators hypothesize that cortisol concentrations are higher, appetite sensations are increased (i.e. increased global appetite score) and food cravings are more prevalent in women of the energy-restriction-plus-CDR group than in women of the energy-restriction-without-CDR group after the 4-week intervention. They also hypothesize that perceived stress is higher and food cravings are more prevalent in women of the energy-restriction-plus-CDR group than in women of the energy-restriction-without-CDR group at 3-month post intervention. They hypothesize that no significant difference in body weight changes is observed between the two groups and that maternal restriction of their child's eating is higher in the energy-restriction-plus-CDR group than in the energy-restriction-without-CDR group both after the 4-week intervention and at the 3-month follow-up.

DETAILED DESCRIPTION:
It is clear that a large proportion of individuals regain weight following dietary weight loss interventions most likely because of homeostatic and non-homeostatic factors favouring a return to initial energy status. However, studies performed to date have documented these effects in the context of interventions favouring both energy restriction and CDR. Thus, the difference between a state of energy restriction alone and a state of energy restriction combined to CDR on factors regulating energy balance is not known. In order to study this important question appropriately, we need to create a condition of energy restriction without increasing CDR, which can only be achieved with a satiating diet (i.e. well-balanced low energy density diet). This is easier to create in the context of a controlled intervention in which all foods and drinks are provided. We propose to create, in a controlled context, an energy restriction for which subjects will be blinded i.e. they will consume less energy than their energy needs without knowing that they are restrained. Such a design will permit to document for the first time the independent effects of CDR in the context of a reduced calorie diet on factors associated with the regulation of energy balance. The proposed study will also allow exploring the impact of increasing CDR on women's attitude toward their children's eating behaviours. Taken all together, results arising from the proposed study will better position the relevance of developing weight loss approaches not focusing on CDR to favour healthy weight management for women and their family. Data will be collected before and after the 4-week intervention, as well as 3 months after the end of the intervention. In order to appropriately test our hypotheses, we cannot state the real purpose of the study in the informed consent form and women will be told that it is a study about the impact of diet on blood pressure. However, at the end of the study, women will be debriefed and will sign a second informed consent form in which the true purpose of the study will be explained.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women (age between 20 to 50 years) from de Quebec City metropolitan area
* Have at least one child (2 to 19 years) living at home
* Body mass index between 25 and 45 kg/m2
* Stable body weight (+/- 2,5 kg) for at least 3 months before the beginning of the study

Exclusion Criteria:

* Women with endocrine disorders, cardiovascular events and type 2 diabetes
* Women with medication that could affect dependent variables measured (namely medication affecting appetite)
* Smokers
* Women with food allergies or food aversion that could impede compliance to the diet
* Pregnant and lactating women
* Women with psychiatric disorders or eating disorders (e.g. bulimia)

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Appetite sensations | At baseline (t=0) and immediately after the 4-week intervention (t=4 wk)
  Measurements of appetite sensations will be performed following a standardized meal. After a 12-hour overnight fast, each woman will be invited to eat a standardized breakfast (600 kcal) and to rate her appetite sensations according to 4 visual analog scales (ranging from 0 to 150 mm): desire to eat, hunger, fullness, and prospective food consumption. Appetite sensations will be recorded before, immediately after, and at 10, 20, 30, 40, 50, and 60 minutes after the consumption of the standardized breakfast.
Stress (cortisol concentrations and perceived stress) | At baseline (t=0), immediately after the 4-week intervention (t=4 wk), and for the perceived stress also at 3 months (t=3 mo) after the end of the intervention
  Cortisol concentrations will be measured by three samples of morning salivary taken immediately at the time of awakening as well as 15 minutes and 30 minutes thereafter. The Perceived Stress Scale will be used to measure perceived stress.

SECONDARY OUTCOMES:
Eating behaviours | At baseline (t=0), immediately after the 4-week intervention (t=4 wk), and 3 months (t=3 mo) after the end of the intervention
  Food craving (Food craving inventory); Cognitive dietary restraint, disinhibition, and susceptibility to hunger (Three factor eating questionnaire); Restrained eating, external eating and emotional eating (Dutch eating behavior questionnaire); Restraint scale; Women's attitude toward their children's eating behaviours (Child feeding questionnaire).
Dietary intakes | At baseline (t=0), immediately after the 4-week intervention (t=4 wk), and 3 months (t=3 mo) after the end of the intervention
  A web-based self-administered food frequency questionnaire will be completed.
Weight | At baseline (t=0), immediately after the 4-week intervention (t=4 wk), and 3 months (t=3 mo) after the end of the intervention
  Weight will be measured.
Waist circumference | At baseline (t=0), immediately after the 4-week intervention (t=4 wk), and 3 months (t=3 mo) after the end of the intervention
  Waist circumference will be measured.
Hip circumference | At baseline (t=0), immediately after the 4-week intervention (t=4 wk), and 3 months (t=3 mo) after the end of the intervention
  Hip circumference will be measured.
Body mass index | At baseline (t=0), immediately after the 4-week intervention (t=4 wk), and 3 months (t=3 mo) after the end of the intervention
  Body mass index will be calculated from measured height and weight.
Lipid profile | At baseline (t=0) and immediately after the 4-week intervention (t=4 wk)
  Basic lipid profile will be measured.
Fasting glycemia | At baseline (t=0) and immediately after the 4-week intervention (t=4 wk)
  Fasting glycemia will be measured.
Fasting insulinemia | At baseline (t=0) and immediately after the 4-week intervention (t=4 wk)
  Fasting insulinemia will be measured.
Systolic and diastolic blood pressure | At baseline (t=0), immediately after the 4-week intervention (t=4 wk), and 3 months (t=3 mo) after the end of the intervention
  Systolic and diastolic blood pressure will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lemieux, Ph.D., Dt.P, Principal Investigator — Department of food sciences and nutrition / Institute of Nutrition and Functional Foods (INAF), Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Laval University, Québec, Quebec, Canada